CLINICAL TRIAL: NCT03199508
Title: Prospective, Randomized, Controlled, Multicenter Clinical Trial of Voiding Diary for Diagnosis and Treatment for Monosymptomatic Enuresis in Children
Brief Title: Clinical Values of Voiding Diary for Diagnosis and Treatment for Monosymptomatic Enuresis in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mao Jianhua (Other)
Collaborators: Jiangxi Province Children's Hospital (Other); Yuying Children's Hospital of Wenzhou Medical University (Other); Shenzhen Children's Hospital (Other Government); Guangzhou Women and Children's Medical Center (Other); Nanjing Children's Hospital (Other); Soochow University (Other)
Responsible Party: Sponsor-Investigator, Mao Jianhua, Chief Physician, The Children's Hospital of Zhejiang University School of Medicine
Organization: The Children's Hospital of Zhejiang University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Voiding Diary Clinical Trial
Record Dates: First submitted 2017-06-19; First posted 2017-06-27 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Nocturnal Enuresis
Keywords: Nocturnal Enuresis; Voiding Diary
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Intervention Model Description: The investigators use two sets of parallel controls. The experimental group use the 3-day voiding diary and the control group use the 7-day voiding diary.
Who Masked: Participant
Masking Description: According to cluster randomization, several centers use the 3-day voiding diary and the other centers use the 7-day voiding diary. Participants will be randomly assigned and don't know they are in which cluster.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the 3-day voiding diary group (Experimental): The 3-day voiding diary group is as the experimental group in which several centers use the 3-day voiding diary by cluster randomization. The 3-day voiding diary is a medical record which need participants to fill in a table about urine volume for 2 days and 3 nights.
  Interventions: Diagnostic Test: the 3-day voiding diary
- the 7-day voiding diary group (Active Comparator): The 7-day voiding diary group is as the control group in which several centers use the 7-day voiding diary by cluster randomization. The 7-day voiding diary is a medical record which need participants to fill in a table about urine volume and drinking water volume for 4 days and 7 nights. The 3-day voiding diary group is the experimental group in which several centers use the 3-day voiding diary by cluster randomization.
  Interventions: Diagnostic Test: the 7-day voiding diary

INTERVENTIONS:
Diagnostic Test: the 3-day voiding diary — The 3-day voiding diary is a medical record which need participants to fill in a table about urine volume for 2 days and 3 nights.
  Arms: the 3-day voiding diary group
Diagnostic Test: the 7-day voiding diary — The 7-day voiding diary is a medical record which need participants to fill in a table about urine volume and drinking water volume for 4 days and 7 nights.
  Arms: the 7-day voiding diary group

SUMMARY:
Nocturnal enuresis is common problem in children who are from 5 to 18 years old and do not spontaneously urinate at least 2 times a week for more than 3 months. It can lead to major distress for the children and their parents. The investigators hypothesize that the 3-day voiding diary as the same as the 7-day voiding diary could be a diagnostic tool to provide information on the diagnosis and classification of nocturnal enuresis. The purpose of this study is to investigate the reliability and sensitivity of 3-day versus 7-day voiding diary to diagnose nocturnal enuresis.

DETAILED DESCRIPTION:
During the first visit to a doctor, a questionnaire about nocturnal enuresis will be filled in and additional tests will be done according to the standard procedure to screen out who have monosymptomatic enuresis.Then participants will complete a 3-day voiding diary or a 7-day voiding diary before treatment. During the second visit to a doctor, doctors will diagnose by voiding diary which type of enuresis is present. Participants need to fill in the 3-day or 7-day voiding diary at 1, 3 and 6 months after standard treatment. About 800 patients from 5 to 18 years old will be included in this prospective, randomized, controlled, multi-center and large sample study and will be followed up at the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Children are from 5 to 18 years old and do not spontaneously urinate at least 2 times a week for more than 3 months.
* Monosymptomatic Enuresis (MNE): children are only associated with nocturnal enuresis, not with daytime lower urinary tract symptoms.

Exclusion Criteria:

* Non-Monosymptomatic Enuresis (NMNE):children have day-time symptoms, such as overactive bladder, discoordinated micturition, dysuria, infrequent voiding and so on.
* Children have psychiatric disorder, urinary tract infection, malformations of the urethra, kidney disease and so on.

  3.Children have been previously treated for nocturnal enuresis who use drugs or other therapeutic regimen.

  4.Secondary enuresis: after 6 months of non-enuresis period, children wet the bed again.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Classification accuracy | 1 week
  According to the results of urinating diary, the subtype of primary nocturnal enuresis would be diagnosed and classified in 400 patients with 3-day diary and 400 patients with 7-day diary, respectively. Then the difference in results of classification accuracy can be evaluated in patients with 3-day diary, compared with 7-day diary which is the golden standard for classification of the subtype of primary nocturnal enuresis.

SECONDARY OUTCOMES:
The compliance rate of two type of urinating diary | 1 month
  The recovery rate would be evaluated when the 3-day diary and 7-day diary were collected in all patients. The compliance rate of two type of urinating diary was evaluated by the recovery rate of diary between 3-day diary and 7-day diary.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, professor, Study Chair — Department of Nephrology, Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- The Children Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaneko K. Treatment for nocturnal enuresis: the current state in Japan. Pediatr Int. 2012 Feb;54(1):8-13. doi: 10.1111/j.1442-200X.2011.03554.x. PMID 22222057
- [Background] Neveus T, Eggert P, Evans J, Macedo A, Rittig S, Tekgul S, Vande Walle J, Yeung CK, Robson L; International Children's Continence Society. Evaluation of and treatment for monosymptomatic enuresis: a standardization document from the International Children's Continence Society. J Urol. 2010 Feb;183(2):441-7. doi: 10.1016/j.juro.2009.10.043. Epub 2009 Dec 14. PMID 20006865
- [Background] Hansen MN, Rittig S, Siggaard C, Kamperis K, Hvistendahl G, Schaumburg HL, Schmidt F, Rawashdeh Y, Djurhuus JC. Intra-individual variability in nighttime urine production and functional bladder capacity estimated by home recordings in patients with nocturnal enuresis. J Urol. 2001 Dec;166(6):2452-5. PMID 11696810
- [Background] Schultz-Lampel D, Steuber C, Hoyer PF, Bachmann CJ, Marschall-Kehrel D, Bachmann H. Urinary incontinence in children. Dtsch Arztebl Int. 2011 Sep;108(37):613-20. doi: 10.3238/arztebl.2011.0613. Epub 2011 Sep 16. PMID 21977217
- See also: Children's monosymptomatic enuresis therapeutic regimen in China — http://kreader.cnki.net/Kreader/CatalogViewPage.aspx?dbCode=CJFD&filename=LCAK201410027&tablename=CJFD2014&compose=&first=1&uid=WEEvREcwSlJHSldRa1FhdXNXYXJwZDB6b0pXbHV0Wkx3VFNDUGI5VXpFQT0=$9A4hF_YAuvQ5obgVAqNKPCYcEjKensW4ggI8Fm4gTkoUKaID8j8gFw!!